CLINICAL TRIAL: NCT05111106
Title: Experience With Symfony Extended Depth of Focus (EDOF) IOL: A Retrospective Chart Review
Brief Title: Symfony Intraocular Lens Retrospective Chart Review
Status: Completed | Type: Observational
Sponsor: Austin Eye (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, John Odette, John Odette, MD, Austin Eye
Other Study IDs: AEJO-2018-Symfony
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Cataract
Keywords: Cataract surgery; Glaucoma; Retinopathy; Intraocular Lens
MeSH Terms: conditions — Cataract; Glaucoma; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Non-Pathology Eyes: Cataract Surgery with implantation of Symfony IOL in eyes without pre-existing pathology..
  Interventions: Device: Symfony IOL
- Glaucoma Eyes: Cataract Surgery with implantation of Symfony IOL with pre-existing glaucoma.
  Interventions: Device: Symfony IOL
- Retinopathy Eyes: Cataract Surgery with implantation of Symfony IOL in eyes with pre-existing retinal pathology..
  Interventions: Device: Symfony IOL

INTERVENTIONS:
Device: Symfony IOL — Implantation of Intraocular lens with extended depth of focus.

SUMMARY:
Retrospective chart review of patients with pre-existing ocular pathology who underwent cataract surgery with implantation of the Symfony IOL.

DETAILED DESCRIPTION:
This was a retrospective chart review conducted at a single US clinical site. Chart review was conducted by John Odette, MD and research assistants. Eligible charts were identified via a clinic database search of cataract surgeries with IOL implantation of the Symfony IOL during the stated date range. Eligible charts included those of patients 18 to 90 years of age who underwent Femto Laser Assisted Cataract Surgery (FLACS) with implantation of a Symfony IOL. Charts were excluded for lack of postoperative follow-up or if Symfony IOL was not implanted. All qualifying patient charts were examined and further classified into 2 groups: (1) eyes with glaucoma; and 2) eyes without glaucoma. Visual acuity was evaluated for patients who underwent cataract surgery with implantation of the Symfony IOL from 09/1/2016 to 05/31/2018. Postoperative evaluations at Month 2 included mean monocular uncorrected visual acuity at near (UNVA) at 40 cm, far distance (UDVA) at 20 ft, and with best correction (CDVA). Outcomes were also compared for toric IOLs versus spherical IOL.

ELIGIBILITY:
Inclusion Criteria:

* :Phacoemulsification cataract surgery with a Symfony IOL.

Exclusion Criteria:

* : Eyes not implanted with a Symfony IOL or unstable refractive results at final post-operative visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-90 years old) in need of cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Monocular uncorrected near visual acuity | 2 months
  handheld near card (Jaeger scale)

SECONDARY OUTCOMES:
Monocular best corrected distance visual acuity | 2 months
  Snellen Chart at 20 feet

CONTACTS AND LOCATIONS:
Overall Officials: John Odette, Principal Investigator — Austin Eye Center

IPD SHARING:
Plan to Share IPD: No